CLINICAL TRIAL: NCT04625374
Title: Prevalence of Chronic Pain After an Emergency Department Visit for Severe Acute Pain and Influence of the Analgesia Initially Used
Brief Title: Prevalence of Chronic Pain After an Emergency Department Visit for Severe Acute Pain
Acronym: CHROPAIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.293; 2020-A02317-32 (Other: ID RCB)
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: EMERGENCY MEDICINE
Keywords: prevalence chronic pain; emergency department; severe acute pain; initial analgesia
MeSH Terms: conditions — Emergencies; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective for investigators is to determine the prevalence of moderate to severe chronic pain in the adult population 6 months after consultation in the emergency department for acute pain (less than 7 days old) and severe pain assessed at admission and defined as greater than or equal to 6/10 by the numerical pain scale.

DETAILED DESCRIPTION:
The presence of pain is the most frequent reason for a patient to visit the emergency department. the investigators know that severe acute pain can be a risk factor for developing chronic pain.

Chronic pain is a symptom, devoid of biological utility, that persists despite the absence of nociceptive stimulus, even after a reasonable period of time that would have allowed the tissue lesion to heal. It is therefore a public health problem with a negative impact on patients' lives.

Chronic pain has been studied in anesthesia and surgery in recent years. In 2006, a study showed the appearance of chronic pain (incidence between 10-50%) in patients who had undergone routine surgery. On the other hand, few studies have looked at the occurrence of chronic pain in patients who came to the emergency department for acute pain.

It is in this context that the investigators find it relevant to assess the prevalence of moderate to severe chronic pain after an emergency department consultation for severe acute pain.

The physiological mechanisms of pain are better identified and the activation of N-methyl-D-aspartate (NMDA) receptors contributes to the onset of hyperalgesia. These receptors are activated under certain conditions, such as during intense and prolonged pain or exposure to high doses of opioids. In addition, the hyperalgesic effect of opioids is known and widely described in the literature. Finally, in the perioperative period, it is now accepted that the administration of a low dose of ketamine can combat these hyperalgesic effects thanks to its NMDA receptor inhibitory action. This effect may have an impact on pain at six months after surgery.

On the basis of these data, it seems relevant to question the prevalence of chronic pain in the course of an emergency department consultation, all the more so in patients with severe initial pain, in whom there is an initial indication for morphine titration, based on the recommendations of the French Society of Emergency Medicine (SFMU).

In addition, the investigators need to question the effects of initial analgesia administered in the emergency department for patients with severe acute pain. Is there a link between the use of certain molecules or the combination of molecules on the onset of chronic pain?

ELIGIBILITY:
Inclusion Criteria:

* To have consulted in the emergency department between 4 to 5 months before reading the files to be contacted 6 months after the consultation in the emergency department;
* Initial pain ≥6 on the Numerical Pain Scale ;
* Acute pain that has been evolving for less than 7 days.
* No oral opposition of the subject required during the phone call

Exclusion Criteria:

* Patient who has undergone surgery in the direct course or within one month of the emergency department visit;
* Patient with suspected or confirmed coronary chest pain at the time of discharge from the emergency department;
* Patient with a mental disability;
* Patient dead;
* Patient who is deaf or hard of hearing;
* Patient who does not speak French or does not live in France
* Patient whose medical history was noted in the file as being impossible due to communication problems;
* Patient who left the emergency department before the end of medical care;
* Patient consulting for acutization of chronic pain;
* Patient during pregnancy;
* Patient consulting for a recent complication of care (within the month), surgical or other;
* Patient taking daily analgesic treatments in the last 2 months;
* Patient known to be dependent on opioids or treated with substitution therapy;
* Homeless patient;
* Patient who has been injured in the course of an assault or violence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who have consulted in the emergency department between 4 to 5 months before reading the files to be contacted 6 months after the consultation in the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Determine prevalence of moderate to severe chronic pain in adult population 6 months after consultation in the emergency department for acute pain (less than 7 days old) and severe pain assessed at admission (defined ≥6/10 by the numerical pain scale) | 6 month
  The main judgment criteria is the presence of chronic pain, related to the pain that motivated the emergency department visit 6 months earlier, moderate to severe defined as pain evolving since the emergency department visit (6 months), experienced at least 2 times per week, and of intensity ≥ 4 on a numerical pain scale during the patient's last painful experience.

SECONDARY OUTCOMES:
To compare the prevalence of chronic pain in patients who initially consulted for pain of traumatic or non-traumatic origin. | 6 month
  Compare the prevalence of moderate to severe chronic pain (defined in the primary end point ≥4/10) in the group of patients who initially consulted for pain from traumatic and nontraumatic causes. Traumatic pain is defined as pain related to a traumatic mechanism less than 1 week old.
Evaluate whether there is an association between the prevalence of chronic pain at 6 months and pain management in use of analgesic, which molecule when the patient goes to the emergency department ; | 6 month
  Association between the prevalence of chronic pain and pain management in the emergency department at analgesic treatment used per molecule
Evaluate whether there is an association between the prevalence of chronic pain at 6 months and pain management in use of analgesic at which dose when the patient goes to the emergency department ; | 6 month
  Association between the prevalence of chronic pain and pain management in the emergency department at the total dose administered to the emergency department
Evaluate whether there is an association between the prevalence of chronic pain at 6 months and pain management at the performance of a locoregional anaesthesia when the patient goes to the emergency department ; | 6 month
  Association between the prevalence of chronic pain and pain management in the emergency department in the realization of a locoregional anaesthesia
Evaluate whether there is an association between the prevalence of chronic pain at 6 months and pain management at the performance of sedation when the patient goes to the emergency department ; | 6 month
  Association between the prevalence of chronic pain and pain management in the emergency department in the performance of procedural sedation
If patients with chronic pain at 6 months reconstructed more often than patients without chronic pain | 6 month
  We will assess whether patients with chronic pain at 6 months reconstruct more often than patients without chronic pain by asking them whether or not they consulted a list of medical specialists, paramedics or did other tests.
The type, characteristics and impact of pain at 6 months after admission to the emergency department. | 6 month
  Brief Pain Inventory Short Form (BPI-SF) questionnaire, 6 months after their visit to the emergency department.
Neuropathic characteristics of pain at 6 months | 6 month
  The neuropathic characteristics of pain will be characterized by the DN-4 questionnaire
Quality of life 6 months after admission to the emergency department | 6 month
  The SF-12 questionnaire will assess quality of life 6 months after admission to the emergency department
Analgesic treatment at 6 months. | 6 month
  Analgesic treatment at 6 months will be evaluated by asking the patient his usual analgesic treatment by class of molecule

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Pellegrin, Bordeaux
  - Grenoble Alpes University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No